CLINICAL TRIAL: NCT03015987
Title: The Effect of Diode Laser Activated Irrigation Versus Ultrasonic Activated Irrigation on Post-Operative Pain in Single Visit Endodontic Treatment of Asymptomatic Necrotic Teeth: A Randomized Controlled Trial
Brief Title: Effect of Diode Laser Activated Irrigation Versus Ultrasonic on Post-Operative Pain in Single Visit of Necrotic Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, zeinab mostafa omar, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: laser_ultrasonic
Record Dates: First submitted 2017-01-04; First posted 2017-01-10 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Necrosis
Keywords: Diode laser; asymptomatic pulp; Laser activated irrigation; continuous ultrasonic activation; post obturation pain
MeSH Terms: conditions — Necrosis | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- diode laser activated irrigation (Experimental): Laser-activated irrigation (LAI) has been introduced as a powerful method enhancing irrigant action; The laser radiation produces transient cavitation in the liquid through optical breakdown by strong absorption of the laser energy. The high-power diode laser has been tested in several areas of dentistry such as bleaching, depigmentation and gingivectomy, with promising results in dentinal disinfection. The diode laser has proved to be a resource worth testing, because of the it's properties and its low cost and availability in comparison to most lasers used in endodontics.
  Interventions: Other: diode laser activated irrigation
- ultrasonic activated irrigation (Active Comparator): ultrasonics have been developed to improve the penetration and effectiveness of irrigation in peripheral areas of the root canal space. The efficiency of sonic and ultrasonic devices is based on the creation of hydrodynamic phenomenon in well-shaped canals filled with an irrigant.
  Such active root canal irrigation has been shown to facilitate the disruption of biofilms and make the cell membrane of bacteria more permeable to NaOCl.
  Interventions: Other: diode laser activated irrigation

INTERVENTIONS:
Other: diode laser activated irrigation — diode laser became the most common and affordable type of laser used in endodontics for many uses , its disinfection effect is an important issue which not discussed in clinical trial before , So this study is assigned to study that
  Other Names: diode laser

SUMMARY:
the investigator intended to study the effect of laser versus ultrasonic in activation of irrigation in post operative pain of patients have a symptomatic necrotic teeth

DETAILED DESCRIPTION:
the investigator will choose from patients entering clinic of endodontics in faculty of oral and dental medicine Cairo university who are eligible to the criteria.

After the patients is found eligible,the patients will be randomly assigned to either the control (ultrasonic activated irrigation )or to the intervention ( diode laser activated irrigation) treatment done in both in single visit.

At the end of treatment, patients will be asked to record post operative pain by NRS .

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic necrotic single rooted single canal teeth with or without chronic periradicular lesion.
* Teeth with mature root
* Teeth without calcified root canals
* Teeth without root caries
* Teeth without internal or external root resorption
* Teeth with no sign of crack formation
* Teeth without anatomic abnormalities

Exclusion Criteria:

* Pregnant or lactating females
* Teeth with vital pulp
* Non- restorable teeth
* Medically compromised patients
* Patients with facial swelling or acute infection.
* Previously endodontically treated teeth
* periodontally affected teeth

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-02; Primary Completion 2018-01 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
post operative pain | up to 1 week
  intensity of post operative pain will be measured using a numerical rating (NRS)scale

CONTACTS AND LOCATIONS:
Overall Officials: Ghada A Eid, Professor, Study Chair — Department of endodontics -Faculty of Oral and Dental Medicine-Cairo university; Hanaa M El shinawy, Researcher professor, Study Director — Surgery &oral medicine department -National Research Institute-Cairo University; Zeinab M Omar, Student, Principal Investigator — Department of endodontics -Faculty of Oral and Dental Medicine-Cairo university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1-Sathorn C, Parashos P, Messer H. The prevalence of postoperative pain and flare-up in single- and multiple-visit endodontic treatment: a systematic review. Int Endod J 2008; 41:91-9. 2-.Ng YL, Glennon JP, Setchell DJ. Prevalence of and factors affecting post. obturation pain in patients undergoing root canal treatment. Int Endod J 2004;37:381-91. 3-Peters OA. Current challenges and concepts in the preparation of root canal systems a review. J Endod 2004; 30:559-67. 4- Gu L, Kim JR, Ling J. Review of contemporary irrigant agitation techniques and devices. J Endod 2009; 35:791-804.